CLINICAL TRIAL: NCT06891963
Title: Transcutaneous Electrical Nerve Stimulation Versus Dry Needling in Non Specific Chronic Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Galal Mohamed Soliman, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003910
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Non Specific Chronic Neck Pain
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture-like TENS + Conventional treatment (Experimental): This group will receive acupuncture like TENS with conventional treatment for 4 weeks.
  Interventions: Other: Acupuncture-like TENS; Other: Conventional treatment
- Dry needling + Conventional treatment (Experimental): This group will receive dry needling with conventional treatment for 4 weeks.
  Interventions: Other: Dry needling; Other: Conventional treatment
- Conventional treatment (Active Comparator): This group will receive conventional treatment for 4 weeks.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Acupuncture-like TENS — The first experimental group will receive 20-minute sessions of TENS, where participants adjust the amplitude to achieve strong muscle twitching beneath the electrodes at an intensity below the pain threshold. Acupuncture-like TENS uses high-frequency pulsed currents at two trains per second with an internal pulse frequency of 100 pps. The pulse pattern is set to "burst," with an asymmetrical biphasic waveform and a pulse duration of 200 µs. Minor fluctuations in pulse rate between 100 and 104 pps were noted using a cathode ray oscilloscope before the experiment.
  Arms: Acupuncture-like TENS + Conventional treatment
Other: Dry needling — The second experimental group will receive 20-minute sessions of dry needling. Patients will be positioned in a prone, relaxed position, and the overlying skin will be cleaned with alcohol. The muscle will be palpated to locate the trigger point (MTrP), with the muscle grasped between the thumb, index, and middle fingers. A solid filiform needle within a guide tube will be inserted into the MTrP using a tapping motion at an oblique angle. The upper trapezius muscle will be palpated for trigger points, with needle insertion depths ranging from 10-15mm. After obtaining a local twitch response, the needle will be moved vertically 3-5mm until no more twitch responses occur. This group will also receive 20 minutes of conventional physical therapy.
  Arms: Dry needling + Conventional treatment
Other: Conventional treatment — All participants in the three groups will receive conventional treatment in the form of hot pack treatment followed by active range of movement (AROM) exercises. A hot pack will be placed on the patients cervical, paraspinal, and upper thoracic areas (including the upper trapezius muscle with aMTrP) for 20 minutes. This will be followed by AROM exercise for cervical spine joints. Participants were asked to actively flex the neck so that the head dropped toward the contralateral trapezius muscles. Patients then rotated the head toward ipsilateral side. This exercise will be repeated five times.

SUMMARY:
This study aims to compare between the effectiveness of Acupuncture-Like Transcutaneous Electrical Nerve Stimulation (Acupuncture-like TENS) and dry needling on pain intensity, Pressure pain threshold (PPT) of upper trapezius myofascial trigger points, neck range of motion, and neck function in patients with non specific chronic neck pain.

DETAILED DESCRIPTION:
The incidence of myofascial trigger points (MTrPs) has been found to vary from 30% to 95% of people who have presented to pain treatment clinics. MPS is common and causes much disability and inability to work so that affect the economy and productivity of workers and employees. According to a previous study, physiotherapy is the most common method used to apply non-invasive techniques and may include the use of modalities for pain relief such as manual therapy, bracing, exercise, Electrical stimulation, kinesio tape, and ultrasound therapy and activity modification. Physiotherapy treatment is recommended to reduce pain, to restore range of motion, function and to strength and stabilize the spine .Trigger points may be relived through many non-pharmacological techniques such as spray and stretch transcutaneous electrical stimulation, massage and dry needing.

Electrotherapy has been widely used as a hypoalgesic agent, which typically involves transcutaneous nerve stimulation. Another well-known hypoalgesic technique is dry needling.

* Acupuncture-Like Transcutaneous Electrical Nerve Stimulation (Acupuncture-like TENS): Acupuncture-like TENS
* Acupuncture-like or Low frequency/High intensity TENS parameters include a low frequency (usually 1-4Hz), a high intensity (high enough to produce visible muscle contractions) and a long pulse duration (~200μs). Acupuncture-like TENS primarily stimulates the Group III (Aδ) and IV (C) nociceptive fibres and small motor fibres. As the mechanism of pain relief associated with this TENS mode requires afferent signals from muscle receptors, the electrodes should be positioned to produce visible muscle contractions, e.g. over a myotome related to the painful area. The user will therefore experience par aesthesia and muscle contraction (twitching type) with this mode. As muscle contractions occur, additional sensory information is carried from the muscle spindle via muscle afferents. This mode of TENS is believed to operate primarily through the release of endogenous opioids via the descending pain suppression system; therefore, there is a relatively longer onset to analgesia but the analgesia typically lasts longer with this mode than with Conventional TENS.

Dry needling (DN) uses a fine, solid needle and is also known as intramuscular stimulation clinical and scientific interest in DN has grown exponentially and various treatment effects are being credited to DN, such as: decreased pain and muscle tension, improved range of motion, muscle strength and coordination.

Although there are many previous studies on the effect of transcutaneous electrical nerve stimulation and dry needling on upper trapezius trigger points, there is no study comparing the therapeutic efficacy between them. However, till now no study compared the therapeutic potential of both modalities. So, this study will be conducted to compare between the effect of transcutaneous electrical nerve stimulation and dry needling in upper trapezius myofascial trigger point.

ELIGIBILITY:
Inclusion Criteria:

Having at least 1 active trigger point in upper trapezius muscles will use a recommended diagnostic criterion to find active MTrPs which is:

* The presence of a palpable taut band in the skeletal muscle.
* The presence of a hypersensitive spot in the taut band.
* Local twitch response provoked by snapping palpation.
* Production of a typical referred pain pattern in response to the compression of tender spots.
* Spontaneous presence of the typical referred pain pattern.
* Duration of symptoms of acute stage (2-4) weeks.
* Age between (20-40) years.
* Having a normal neurological examination result .

Exclusion Criteria:

* Existence of cervical disc hernia, advanced cervical osteoarthritis, radiculopathy, or myelopathy.
* Having trigger point injection or physical therapy in the last 6 months.
* Having a rheumatologic disease, such as fibromyalgia, rheumatoid arthritis, or a hormonal disease, such as hypothyroidism, hyperthyroidism or hyperparathyroidism.
* Existence of kyphosis, scoliosis, forward head posture or cervicogenic headache.
* History of spine surgery.
* Having a cardiovascular problem.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of neck pain intensity | 4 weeks
  The Visual Analogue Scale (VAS) will be used to evaluate pain intensity. It is a horizontal line whose length is 10 cm; its left end (zero) indicates no pain, while its right end (ten) reveals the worst imaginable pain. Each subject will be in relaxed position and will be asked to mark the point on the line that exactly corresponded to his/her pain.
Assessment of pressure pain threshold (PPT) | 4 weeks
  The pressure pain threshold (PPT) will be assessed by positioning the tip of the algometer on the trigger point and increasing the pressure by 1 kg per second. When the patient indicates discomfort, the pressure value will be recorded in kg/cm. The procedure will be repeated three times at 60 s intervals, and the mean pressure value will be recorded as the PPT.

SECONDARY OUTCOMES:
Measurement of cervical flexion range of motion (ROM) | 4 weeks
  It will be measured for all participants in the three groups pre- and post-treatment, using the CROM device. Each participant will asked to perform cervical flexion three times and the mean value will be recorded.
Measurement of cervical extension ROM | 4 weeks
  It will be measured for all participants in the three groups pre- and post-treatment, using the CROM device. Each participant will asked to perform cervical extension three times and the mean value will be recorded.
Measurement of cervical lateral flexion to the right ROM | 4 weeks
  It will be measured for all participants in the three groups pre- and post-treatment, using the CROM device. Each participant will asked to perform cervical lateral flexion to the right three times and the mean value will be recorded.
Measurement of cervical lateral flexion to the left ROM | 4 weeks
  It will be measured for all participants in the three groups pre- and post-treatment, using the CROM device. Each participant will asked to perform cervical lateral flexion to the left three times and the mean value will be recorded.
Measurement of cervical rotation to the right ROM | 4 weeks
  It will be measured for all participants in the three groups pre- and post-treatment, using the CROM device. Each participant will asked to perform cervical rotation to the right three times and the mean value will be recorded.
Measurement of cervical rotation to the left ROM | 4 weeks
  It will be measured for all participants in the three groups pre- and post-treatment, using the CROM device. Each participant will asked to perform cervical rotation to the left three times and the mean value will be recorded.
Assessment of neck function | 4 weeks
  The Neck Disability Index (NDI) will be used to assess functional status for all participants in the three groups before and after treatment. The NDI is a 10-item questionnaire assessing personal care, pain, reading, lifting, concentration, headaches, work, driving, sleeping, and recreation. Each item is scored from 0 (no disability) to 5 (total disability), with a maximum possible score of 50. Participants will select the answer that best describes their neck function. Total scores are categorized as follows: 0-4 (no disability), 5-14 (mild disability), 15-24 (moderate disability), 25-34 (severe disability), and 35+ (complete disability).

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Abdel Latif Abdel Raoof, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Zagazig general hospital, Zagazig, Egypt